CLINICAL TRIAL: NCT05682625
Title: Understanding COVID-19 Vaccine Immunity in Tissue and Blood
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty with enrollment
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Associate professor, Stanford University
Other Study IDs: IRB-67705; 1U19AI167903-01 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19 (Coronavirus Disease 2019)
Keywords: Immunity; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lymph node biopsy and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adults who are receiving a COVID-19 vaccine
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this study is to understand the effects of COVID-19 vaccines on the immune system and how the COVID-19 vaccines provide protection and induce long term memory. Adults who are receiving a COVID-19 vaccine will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18yrs old and higher who are receiving a COVID-19 vaccine

Exclusion Criteria:

* Pregnancy
* Patients with contraindications for lymph node biopsy
* Active cancer
* Current use of immunosuppression drugs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (18 years and older) receiving a COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Testing immune response to the COVID-19 vaccine over time | 1 day
Testing immune response to the COVID-19 vaccine over time | 7 days
Testing immune response to the COVID-19 vaccine over time | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: R. Sharon Chinthrajah, MD, Principal Investigator — Stanford University, Sean N. Parker Center for Allergy and Asthma Research
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No